CLINICAL TRIAL: NCT05561309
Title: A Phase Ⅱ Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Single Injection Adductor Canal Block With HR18034 for Postoperative Pain Management
Brief Title: Phase Ⅱ Study of Adductor Canal Block With HR18034 for Postsurgical Pain Management
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HR18034-201
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: HR18034 compared with active comparator
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dose 1 (Experimental): Experimental: HR18034 190mg (10ml)
  Intervention: Drug: HR18034
  Active Comparator: Ropivacaine Hydrochloride Injection
  Ropivacaine Hydrochloride Injection 50mg (10mL)
  Intervention: Drug: Ropivacaine Hydrochloride Injection
  Interventions: Drug: HR18034;Ropivacaine Hydrochloride Injection
- dose 2 (Experimental): Experimental: HR18034 285mg (15ml)
  Intervention: Drug: HR18034
  Active Comparator: Ropivacaine Hydrochloride Injection
  Ropivacaine Hydrochloride Injection 75mg (15mL)
  Intervention: Drug: Ropivacaine Hydrochloride Injection
  Interventions: Drug: HR18034;Ropivacaine Hydrochloride Injection
- dose 3 (Experimental): Experimental:HR18034 380mg (20ml)
  Intervention: Drug: HR18034
  Active Comparator: Ropivacaine Hydrochloride Injection
  Ropivacaine Hydrochloride Injection 100mg (20mL)
  Intervention: Drug: Ropivacaine Hydrochloride Injection
  Interventions: Drug: HR18034;Ropivacaine Hydrochloride Injection

INTERVENTIONS:
Drug: HR18034;Ropivacaine Hydrochloride Injection — Drug: HR18034
  Drug: Ropivacaine Hydrochloride Injection
  Local nerve block of Ropivacaine Hydrochloride Injection to produce anesthesia for surgery and analgesia in postoperative pain management.
  Other Name: Ropivacaine Hydrochloride Injection, 0.5% Injectable Solution

SUMMARY:
Phase Ⅱ, randomized, double-blind, comparator-controlled study to evaluate the efficacy, safety and pharmacokinetics of single injection adductor canal block with HR18034 for postoperative pain management compared with ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Scheduled to undergo primary unilateral total knee arthroplasty under general anesthesia.
3. Male or female，aged 18-75 years inclusive
4. Body mass index (BMI) 18-28 kg/m2 inclusive
5. American Society of Anesthesiologists (ASA) Physical Status Classification Ⅰ~Ⅱ

Exclusion Criteria:

1. Subjects with deformity of the involving operative limb, or other neuropathy
2. Subjects with a history of new myocardial infarction or unstable angina within 6 months prior to randomization;
3. Subjects with a history of ischemic stroke or transient ischemic attack (TIA)
4. Subjects with a history of mental system diseases and cognitive dysfunction
5. Combination of other pain conditions that may affect postoperative pain assessment
6. Persistent or recurrent nausea and/or vomiting due to other etiologies, including, but not limited to gastric outlet obstruction, hypercalcemia, or active peptic ulcer
7. Subjects with a history of deep vein thrombosis-related disease
8. Clinically significant abnormal clinical laboratory test value
9. Allergic to a drug ingredient or component
10. Use of any of medications, which affect drug metabolism or analgesia evaluation, within 5 half-lives or as specified prior to the study surgical procedure
11. History of alcohol abuse or prescription and/or illicit drug abuse
12. Subjects with special diets (including tobacco, grapefruit and caffeine)
13. Pregnant or nursing women
14. No birth control during the specified period of time
15. Participated in clinical trials of other drugs (received experimental drugs)
16. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
AUC0-72 of the NRS-R pain intensity scores. | 0 to 72 hours
  AUC of NRS pain intensity scores at rest (NRS-R) through 72 hours after the beginning of study drug administration.

SECONDARY OUTCOMES:
AUC of the NRS-R pain intensity scores. | 0-24, 0-48 hours
  AUC of NRS pain intensity scores at rest (NRS-R) for time periods 0-24, 0-48 hours.
AUC of the NRS-A pain intensity scores. | 0-24, 0-48, 0-72 hours
  AUC of NRS pain intensity scores at activity (NRS-A) for time periods 0-24, 0-48, 0-72 hours.
Pain intensity assessed using an 11-point NRS ranging. | Baseline till 72 hours after the beginning of study drug administration
  11-point Numercal Rating Scale ranging from a score of 0 to 10. Pain-free defined as an NRS of 0 or 1. Worst imaginable pain defined as an NRS of 10
Proportion of subjects who used no rescue opioid analgesic. | 0-24, 24-48, 48-72, 0-72 hours
  Proportion of subjects who used no rescue opioid analgesic through 0-24, 24-48, 48-72 and 0-72 hours after the beginning of study drug administration.
Total rescue analgesic consumption. | 0-24, 24-48, 48-72, 0-72 hours
  Total rescue analgesic consumption through 0-24, 24-48, 48-72 and 0-72 hours after the beginning of study drug administration.
Time to the first postoperative use of rescue opioid analgesics. | 0-72hours
  Time to the first postoperative use of rescue opioid analgesics 0-72 hours after the beginning of study drug administration.
Quadriceps muscle strength score. | Baseline till 72 hours after the beginning of study drug administration
  Quadriceps muscle strength score at 6, 8, 12, 16, 20, 24, 36, 48 and 72 hours.
Subjects' satisfaction rating | 72 hours
  Subjects' satisfaction rating with postsurgical pain control at 72 hours.
Investigators' satisfaction rating | 72 hours
  Investigators' satisfaction rating with postsurgical pain control at 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguan People's Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided